CLINICAL TRIAL: NCT03838913
Title: Classification of Mutation Characteristics by Whole-Exome Sequencing (WES) in Intraductal Neoplasms of the Bile Duct (IPNB) Patients
Brief Title: Whole-Exome Sequencing (WES) of Intraductal Neoplasms of the Bile Duct (IPNB)
Acronym: WESIPNB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fujian Provincial Hospital (Other)
Collaborators: Fujian Medical University Union Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Yaodong Wang, Director of Dept. Hepatobiliary Surgery, Fujian Provincial Hospital
Other Study IDs: Fujian Provincial Hospital
Record Dates: First submitted 2019-01-13; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Bile Duct Neoplasms; Intraductal Papillary Mucinous Neoplasm
Keywords: Whole-exome Sequencing; intraductal papillary neoplasms of the bile duct; mutation characteristics
MeSH Terms: conditions — Bile Duct Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IPNB: intraductal papillary neoplasm of the bile duct

SUMMARY:
Intraductal papillary neoplasm of the bile duct (IPNB) is a distinct type of biliary tumor characterised with delicate fibrovascular stalks (papillary of villous) covered at biliary epithelium. The typical pathologic feature is dramatical dilation of affected bile ducts due to obstruction by mucin production. IPNB has a better prognosis than bile duct carcinoma, but the current proposed entity contains multiple definitions or categories, thus confused in pathology.

Although mutations of several genes on IPNBs (such as GNAS, KRAS, APC, CTNNB1, and RNF43) identified in previous studies, there is still an unification at gene expression signature.

This research trial will use whole exome sequencing and subsequent bioinformatic analysis in finding causative mutations in deoxyribonucleic acid (DNA) samples from IPNBs patients.

DETAILED DESCRIPTION:
Using production-scale platform, this study will carry out whole exome sequencing from archival (FFPE) material to Identification and classification of significantly mutated genes, determine the somatic genomic alterations that may be relevant to the development or treatment of cancer, establish classification of IPNBs gene mutation signature. Next, analysis of gene mutation signature and IPNBs clinicopathologic outcomes, including the association between pathologic type, long-term oncological outcomes and gene mutation signature. Last, the determination of involved signal pathways at IPNB patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IPNBs
* ECOG Performance status of 0, 1, or 2
* Adequate liver function, bilirubin < 1.5 times ULN, ALT or AST < 2.5 times ULN
* Adequate renal function: creatinine < 1.8
* Must be at least 18

Exclusion Criteria:

* Diagnosis of hepatic mucinous cystadenoma (MCN)
* Complicated with other Malignancy
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 cases
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of novel genetic contributors to IPNBs | 1 year
  Novel genetic abnormalities that are found to be associated with IPNBs via production-scale platform for whole exome sequencing from archival (FFPE) material. The tumor and normal specimens will be obtained from patients with IPNBs who are receiving treatment at Fujian Provincial Hospital, Fujian Medical University Union Hospital and First affiliated Hospital of Fujian Medical University.
Validation of WES outcomes | 1 year
  To precise determination of mutation signature of WES results by Sanger Sequencing.
Determination of involved signal pathways | 1 year
  To predict and verify the involved signal pathways by bioinformatics

CONTACTS AND LOCATIONS:
Overall Officials: Yaodong Wang, Prof, Principal Investigator — Fujian Provincial Hospital
Locations (1):
- Yaodong Wang, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No